CLINICAL TRIAL: NCT01982656
Title: Effects of Massage Technique for Pain, Anxiety, and Delirium Management in ICU Patients With Subarachnoid Hemorrhage
Brief Title: Massage Technique for Pain, Anxiety and Delirium in SAH Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sara E. Hocker, M.D (Other)
Responsible Party: Sponsor-Investigator, Sara E. Hocker, M.D, Principle Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-003346
Record Dates: First submitted 2013-10-16; First posted 2013-11-13 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Subarachnoid Hemorrhage; Anxiety; Pain; Delirium; Sleep
MeSH Terms: conditions — Subarachnoid Hemorrhage; Anxiety Disorders; Pain; Delirium | interventions — Massage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Massage technique (Experimental): In addition to standard medical care and pharmacologic interventions, massage technique for 20 minutes for 5 to 14 days while in the ICU will be provided to help alleviate pain and anxiety in the patient.
  Interventions: Other: Massage
- No intervention (Placebo Comparator): Patients with an aneurysmal subarachnoid hemorrhage will receive standard medical care to include pharmacologic interventions prescribed by the primary physician and nonpharmacologic interventions provided by the bedside RN such as ice or heat to address their pain and anxiety needs.
  Interventions: Other: Massage

INTERVENTIONS:
Other: Massage — twenty minute massage intervention prior to bedtime (1900-2100), to be started after day 3 of admission for a minimum of 5 consecutive days and up to fourteen days. The massage will be conducted by an RN trained in massage technique that is not caring for the patient in a direct nursing role.

SUMMARY:
This research study seeks to explore the effects of massage techniques on pain and anxiety relief among patients with subarachnoid hemorrhages in the ICU setting in comparison to subarachnoid hemorrhagic patients using standard medical therapy. In addition, our aim is to decrease the overall medication use to treat pain and anxiety, and to determine the impact of massage on sleep duration, quality, and breathing. Our goal is to improve and promote comfort during the ICU stay as well as decrease the need for narcotic medication usage.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of aneurysmal subarachnoid hemorrhage

Exclusion Criteria:

* Upper extremity deep vein thrombus
* Active alcohol or drug withdrawal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-12; Primary Completion 2017-12-31 (Actual); Study Completion 2018-02-22 (Actual)

PRIMARY OUTCOMES:
Change in Pain Score | Baseline to 14 days
  Over the course of the intervention period, the primary outcome of decrease in pain will be decreased as compared to the control group. This will be measured using the Pain Scale.

SECONDARY OUTCOMES:
Sleep quantity | 5-14 days

CONTACTS AND LOCATIONS:
Overall Officials: Sara Hocker, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Background] Zolfaghari M, Eybpoosh S, Hazrati M. Effects of therapeutic touch on anxiety, vital signs, and cardiac dysrhythmia in a sample of Iranian women undergoing cardiac catheterization: a quasi-experimental study. J Holist Nurs. 2012 Dec;30(4):225-34. doi: 10.1177/0898010112453325. Epub 2012 Jul 24. PMID 22828950
- [Background] Valiee S, Bassampour SS, Nasrabadi AN, Pouresmaeil Z, Mehran A. Effect of acupressure on preoperative anxiety: a clinical trial. J Perianesth Nurs. 2012 Aug;27(4):259-66. doi: 10.1016/j.jopan.2012.05.003. PMID 22828022
- [Background] Bauer BA, Cutshall SM, Wentworth LJ, Engen D, Messner PK, Wood CM, Brekke KM, Kelly RF, Sundt TM 3rd. Effect of massage therapy on pain, anxiety, and tension after cardiac surgery: a randomized study. Complement Ther Clin Pract. 2010 May;16(2):70-5. doi: 10.1016/j.ctcp.2009.06.012. Epub 2009 Jul 14. PMID 20347836